CLINICAL TRIAL: NCT01279655
Title: The Influence of a tDCS Combined Long-term Motor Training Program on Structural White Matter Changes in the Brain, Functionality and Psychological Outcome Measures in Multiple Sclerosis.
Brief Title: Motor Training and White Matter in Multiple Sclerosis (MS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: KU Leuven (Other); Provinciale Hogeschool Limburg (Other)
Responsible Party: Principal Investigator, Koen Cuypers, Drs, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MECU2012-001
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tDCS and training (Experimental): Transcranial Direct current stimulation (tDCS) is applied together with a bimanual learning task. tDCS is delivered through two gel-sponge electrodes (eldith DC Stimulator, neuroConn GmbH, Ilmenau, Germany) embedded in a saline-soaked solution. tDCS will be applied for 20 min, with a current intensity of 1mA.
  Interventions: Device: tDCS; Behavioral: Bimanual Training
- Control (No Intervention): No intervention is applied
- Sham tDCS + Training (Placebo Comparator): The training consists of a bimanual training task. tDCS is only applied for a few seconds and will than be ramped-down.
  Interventions: Device: tDCS; Behavioral: Bimanual Training

INTERVENTIONS:
Device: tDCS — 20 min, 1mA, 8 weeks (5 days a week, 20 min a day)
  Other Names: eldith, neuroConn, serial 0118
  Arms: Sham tDCS + Training; tDCS and training
Behavioral: Bimanual Training — The training program consisted of a bimanual etch-a-sketch task. By rotating two wheels subjects have to match a line presented on the screen with the cursor. 8 weeks (5 days a week, 20 min a day)
  Arms: Sham tDCS + Training; tDCS and training

SUMMARY:
In the current study the researchers will firstly investigate whether a bimanual coordination training protocol (20 min/day, for 8 consecutive weeks) correlates with changes in white matter architecture and improved upper-limb functionality in patients with multiple sclerosis. Secondly, the researchers predict that motor learning is more efficient when it is combined with anodal transcranial direct current (tDCS) stimulation on the left primary motor cortex.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) scores between 2 and 6.5
* Stable MS (no relapse during the last 3 months before study onset)
* age: between 18 and 68 years

Exclusion Criteria:

* Patients with other pathologies associated with peripheral and/or central sensory dysfunction or under psychotropic or antiepileptic medication.
* Standard TMS/tDCS and MRI exclusion criteria (safety questionnaires)

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Change in White Matter | Baseline, immediately after and 3 weeks after the intervention
  Diffusion Tensor Imaging (DTI) T1 structural scan Fluid-attenuated inversion recovery Scan (FLAIR) Magnetization Transfer Imaging (MTI)

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, immediately after and 3 weeks after the intervention
  Questionnaire
Blood sample | After the end of the study
  BDNF Genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Raf Meesen, Phd, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University (BIOMED), Diepenbeek, Limburg, Belgium